CLINICAL TRIAL: NCT06958796
Title: Exploratory Use of CMV Immunoglobulin in High Risk (D+R-) Transplant Recipients at the End of Antiviral Prophylaxis to Decrease the Risk of Late CMV Infection
Brief Title: Strategic Help With Immunoglobulin to Enhance Protect Against Late Disease (CMV)
Acronym: SHIELD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Camille N. Kotton, MD (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Kamada, Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Camille N. Kotton, MD, Camille N. Kotton, MD, Clinical Director of Transplant Infectious Disease, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024P003592
Record Dates: First submitted 2025-04-18; First posted 2025-05-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cytomegalovirus; Organ Transplant; Kidney Transplant; Complications; Liver Transplant Complications; Simultaneous Liver-Kidney Transplantation; Complications
Keywords: cytomegalovirus; valganciclovir; organ transplant; immunoglobulin; CMV; High Risk CMV

STUDY DESIGN:
Intervention Model Description: This research study will compare CytoGam® used after valganciclovir in D+R- liver, kidney, or liver-kidney transplant recipients to valganciclovir alone. Valganciclovir is used routinely to prevent CMV disease. Qualifying participants are assigned to a study group by chance (like a coin toss) to Arm A, the CytoGam® group or Arm B, the standard of care group. Neither the subject nor the study doctor can choose the study group. Participants will have an equal chance of being assigned to the CytoGam® group.
Masking Description: This is an open label study so both participants and study doctor will know which arm has been assigned; no placebo infusion is planned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: CytoGam® (Experimental): Participants assigned to receive CytoGam® will receive an infusion once a month for three months at their study site. The infusion will be completed over an average of about 4 hours; these three visits will last about 5 hours. During these study staff will review concomitant medications and adverse events. Participants will be asked to have blood taken at infusion visits and 2 weeks after an infusion visit to check the level of CMV DNA in their blood.
  Interventions: Drug: Cytomegalovirus Immune Globulin Intravenous (Human) monthly for three months
- Arm B: Standard of Care (No Intervention): Participants assigned to Arm B, will be asked to complete a telephone call visit once a month. During these visits, a member of study staff will review concomitant medications and adverse events. Participants will be asked to have their blood taken every two weeks to check the level of CMV DNA.

INTERVENTIONS:
Drug: Cytomegalovirus Immune Globulin Intravenous (Human) monthly for three months — The interventional arm will receive Cytomegalovirus Immune Globulin Intravenous (Human) monthly for three months as (150 mg/kg) for 3 consecutive months (Days 0, 28 and 56 +/- 3 days). The non-interventional arm will not receive any intervention.
  Arms: Arm A: CytoGam®

SUMMARY:
This study is being done to find out if administering CytoGam® after the end of standardly prescribed preventive antiviral treatment can help transplant recipients with a high risk for developing late CMV disease after a liver and/or kidney transplant.

DETAILED DESCRIPTION:
This research study is being done to find out if administering CytoGam® after the end of standardly prescribed preventive antiviral treatment can help people with a high risk for developing late CMV disease post-transplant.

Cytomegalovirus (CMV) is a very common virus and in the same family as the viruses that cause herpes, chickenpox, and mononucleosis. Most people become infected with the virus when they come in direct contact with an infected person's bodily fluids. People with a normal immune system who become infected with CMV can have no symptoms or have symptoms similar to the common cold; people with a normal immune system rarely have any major complications from the virus. Once someone is infected with CMV, the virus remains inactive, or dormant, in the body for life; sometimes the virus can become active again and cause symptoms or severe disease, especially in people who are sick or have a weak immune system.

Individuals who receive an organ transplant are more likely to get an active CMV infection because of the medications required to prevent the immune system from attacking the transplanted organ. The immune system might recognize the organ transplant as a threat because it is not made of the same cells as the rest of the body. Anti-rejection medications help to reduce the immune system from attacking and damaging a new organ but also make it harder to fight off CMV and other infections. CMV is one of the most common infections after transplant.

Transplant teams test for CMV when someone is listed for an organ transplant and right before surgery. Both donors and recipients are tested for a CMV antibody which determines if someone has ever been infected with CMV. An antibody is created by the immune system and helps fight dangerous invaders like bacteria, fungus, or a virus, like CMV. People develop an antibody if the virus has been present in their body at any point in their life. CMV is so common that healthy people who test positive for CMV can still be organ donors; about half of all American adults have previous CMV infections.

The transplant team looks at the CMV antibody test results from both a donor and recipient at the time of the transplant surgery to determine the level of possible risk for CMV disease occurring in the recipient. Below is information regarding the level of potential risk to the recipient based on the presence (+) or absence (-) of antibodies. Other factors can influence someone's risk of CMV disease after transplant and can include age (of donor and recipient), other health problems, type and dosage of certain anti-rejection medications taken after transplant, and symptoms of transplant rejection.

Risk Levels Lowest (D-/R-): Neither the donor nor the recipient have been infected with CMV. This match presents the lowest risk of CMV disease to the recipient.

Moderate (D-/R+ or R+/R+): When the recipient is positive for the antibody, they have some immunity, or protection, to the virus so they face a moderate risk for CMV disease regardless of their donor's CMV status. These mismatches present a moderate risk for CMV disease.

Highest (D+/R-): The highest risk for CMV disease occurs when a donor is positive for the antibody, but the recipient is negative. In this situation, the virus is present in the donor's body, but the recipient has no antibodies or immunity/protection against the virus. This mismatch presents the highest risk for CMV disease.

When someone has CMV before transplant, there is a risk the virus will reactivate after transplant when the immune system is suppressed. These patients have some protection against the virus because there are antibodies, or immunity, present in the body which helps reduce the risk for severe CMV disease. If a transplant recipient has never had CMV but receives an organ from someone who had CMV there is no natural protection against the virus and those individuals face the highest risk for CMV disease.

CMV disease may cause flu-like symptoms like fever, chills, fatigue, and muscle aches. CMV can also cause infection in different types of tissues and other types of CMV disease like:

Pneumonia (a lung infection that causes fever, cough, labored breathing) Gastrointestinal disease (indigestion, nausea, vomiting, abdominal pain, bloating, diarrhea) Hepatitis (inflammation of the liver) Central nervous system disease (infection of the brain or spinal cord causing weakness, decreased memory, confusion) Retinitis (inflammation of the retina, a part of the eye, which impact vision) Organ dysfunction-CMV can impact the function of other organs and affect a transplanted organ Organ rejection Death

CMV disease usually occurs in the first few months after transplant when anti-rejection medications are taken in higher doses and the immune system is at its weakest. During this high-risk period, transplant recipients at a moderate or high CMV risk are prescribed an antiviral medication, valganciclovir. Prophylactic, or preventive, treatment with valganciclovir greatly reduces the risk for CMV disease but some recipients still develop late CMV disease, which occurs more than 100 days after transplant. The risk for late CMV disease is highest in individuals who did not have a CMV infection (R-) before transplant but received an organ from someone who had CMV (D+). This mismatch is written as D+R-.

The length of time someone is on prophylactic treatment after organ transplant depends on the type of organ they receive and their risk level. D+R- liver transplant recipients are often prescribed valganciclovir for 3 months while D+R- kidney transplant recipients often take valganciclovir for 6 months. Following valganciclovir treatment, some recipients may have their blood tested every 1 to 2 weeks for 3 months to monitor how much CMV is the body; this test, called a CMV PCR test looks for the DNA of the virus and can help the transplant team assess the recipient's risk for CMV disease, diagnose CMV quickly, and monitor treatment effectiveness and development of antiviral resistance.

This research is being done to explore if the risk of late CMV disease following a D+R- a liver, kidney, or simultaneous liver-kidney transplant can be further reduced with CytoGam® infusions after the standardly prescribed prophylactic antiviral medications.

CytoGam® is an intravenous immunoglobulin or IVIG. Immunoglobulin is another name for an antibody and helps the body fight infection; intravenous immunoglobulin is made with collected antibodies from healthy donors and is like a blood transfusion from donated blood. A CytoGam® infusion delivers immunoglobulin, or antibodies, specific to CMV to help strength the immune system's natural defenses.

CytoGam® is approved by the U.S. Food and Drug Administration (FDA) for the prophylaxis, or prevention, of CMV disease associated with transplantation of kidney, lung, liver pancreas, and heart, but CytoGam® is not approved by the FDA to be administered after antiviral prophylaxis to prevent CMV disease or reduce CMV severity.

ELIGIBILITY:
Inclusion Criteria

* High risk pretransplant CMV donor seropositive/recipient seronegative (D+R-) kidney, liver, or simultaneous liver-kidney (SLK) transplant recipients
* Able to do routine blood testing (normal care for transplant recipients)
* Written informed consent obtained from the subject before any trial-related procedures
* Be ≥18 years and ≤75 years of age at time of consent

Exclusion Criteria

* Any pre-transplant CMV serologic combinations besides CMV D+/R-
* Multi organ transplants (other than simultaneous liver-kidney transplant (SLK) recipients) or prior history of bone marrow or stem cell transplant
* Lung, heart, small bowel, pancreas, or other non-kidney or non-liver transplant recipients
* Transplant recipients treated for rejection within three months before the end of valganciclovir prophylaxis
* Participation in another interventional clinical trial at time of consent or within 30 days prior to study consent
* Transplant recipients with eGFR <30 ml/min/1.73m2 (as they theoretically could be at higher risk for renal impairment with CMV immunoglobulin), poor transplant organ function (i.e. LFTs > twice the upper limit of normal in liver recipients), or who are on dialysis, or plasmapheresis, or who are relisted for transplant, or who might otherwise at risk of complications at the discretion of the local site investigator.
* Those with a history of severe reaction to CMV immunoglobulin (e.g. CytoGam® or similar) or other human immunoglobulin preparations
* Individuals with a history of selective immunoglobulin A deficiency will be excluded, as they may produce antibodies against immunoglobulin A, leading to potential anaphylactic reactions upon receiving blood products containing immunoglobulin A, such as CMV immunoglobulin (e.g. CytoGam® or similar)
* Any history of acute myocardial infarction (within 12 months of screening), clinically significant arrythmia, or clinically significant ECG abnormality in the opinion of the investigator at time of screening
* History of active or latent tuberculosis (except those who have completed a documented regimen for latent TB treatment) or severe pulmonary disease [e.g., severe pulmonary hypertension (WHO class IV)] that in the opinion of the investigator that may preclude their ability to safely tolerate study infusions
* Any history of neurodegenerative disease, including dementia, or stroke with substantial residual disability (modified Rankin score ≥ 3)
* Pregnant or nursing (lactating) women confirmed by human chorionic gonadotropin (hCG) laboratory test.
* Women of childbearing potential unless using a highly effective method of contraception during dosing and for 24 weeks after study treatment. Medically acceptable birth control (contraceptives) includes but are not limited to: surgical sterilization (such as hysterectomy or "tubes tied"), approved hormonal contraceptives (such as birth control pills, patch or ring; Depo-Provera, Depo-Lupron, lmplanon), barrier methods (such as condom or diaphragm), an intrauterine device (IUD), abstinence from sex.
* Any significant history of any treatment nonadherence or any other medical condition that, in the investigator's opinion, would confound the results of the study or put the participant at undue risk
* Subjects who have any of the following laboratory values: eGFR <30 ml/min/1.73m2 ; Hemoglobin <8.0 g/dL; Platelets <50,000 cells/uL; Absolute neutrophil count <1,000 cells/uL; Total bilirubin >2.5 x upper limit of normal; Alanine aminotransferase (ALT) >5 x upper limit of normal; Aspartate aminotransferase (AST)] >5 x upper limit of normal; CMV IgG negative in donor or positive in recipient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Late Clinically Significant CMV Disease | Treatment Phase (Day 0) through End of Study (Day 168)
  Comparison between treatment groups of number of participants with a blood CMV viral load >1000 IU/ml at any point during the treatment phase through end of study
Number of Participants with Adverse Events Related to CMV | Events starting after or increasing in severity following initiation of the Treatment Phase (Day 0) through end of study (Day 168)
  Congregate data of all Adverse Events (including Serious Adverse Events) will be compared between treatment arms. The number and percent of CMV related AEs will be summarized by:
  Organ system impacted Relationship to CMV Severity Deaths
  Those leading to:
  1. Initiation of CMV treatment
  2. Hospitalization due to CMV

SECONDARY OUTCOMES:
Peak CMV DNA Levels | From Enrollment, through the Treatment Phase (Day 0) until the end of study (Day 168)
  Comparison of peak CMV DNA levels (DNAemia/viremia) between treatment groups using either the Wilcoxon rank-sum test or Student's t-test, depending on the distribution of the data; DNA tests will be completed every 2 weeks throughout the trial and reported in IU/ml
Change in CMV DNA Levels Across Study Groups | From Enrollment, through the Treatment Phase (Day 0) until the end of study (Day 168)
  Trend the change and differences in CMV viral loads over time between groups using a mixed-effects model with biweekly CMV DNA test results
Time to First Detectable CMV DNAemia | Treatment Phase (Day 0) through End of Study (Day 168)
  Time to onset of CMV DNAemia/viremia summarized by treatment group measured by week of onset after day 0 (end of valganciclovir prophylaxis)

CONTACTS AND LOCATIONS:
Overall Officials: Camille Kotton, MD, FIDSA, FAST, Principal Investigator — Massachusetts General Hospital; David Wojciechowski, DO, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The two study sites will share IPD using a REDCap database. This will be done under a data use agreement signed by both institutions. Data will not be shared beyond the two study sites.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be shared during and after the study during data analysis. We anticipate the study will start in May 2025 and supporting information will be available for the following three years.
Access Criteria: IPD will be available to the investigators at each institution through the REDCap database.

REFERENCES:
- [Background] Kotton CN, Kumar D, Caliendo AM, Huprikar S, Chou S, Danziger-Isakov L, Humar A; The Transplantation Society International CMV Consensus Group. The Third International Consensus Guidelines on the Management of Cytomegalovirus in Solid-organ Transplantation. Transplantation. 2018 Jun;102(6):900-931. doi: 10.1097/TP.0000000000002191. PMID 29596116
- [Background] Razonable RR, Humar A. Cytomegalovirus in solid organ transplant recipients-Guidelines of the American Society of Transplantation Infectious Diseases Community of Practice. Clin Transplant. 2019 Sep;33(9):e13512. doi: 10.1111/ctr.13512. Epub 2019 Mar 28. PMID 30817026
- [Background] McBride JM, Sheinson D, Jiang J, Lewin-Koh N, Werner BG, Chow JKL, Wu X, Tavel JA, Snydman DR. Correlation of Cytomegalovirus (CMV) Disease Severity and Mortality With CMV Viral Burden in CMV-Seropositive Donor and CMV-Seronegative Solid Organ Transplant Recipients. Open Forum Infect Dis. 2019 Jan 14;6(2):ofz003. doi: 10.1093/ofid/ofz003. eCollection 2019 Feb. PMID 30775403
- [Background] Ljungman P, Chemaly RF, Khawaya F, Alain S, Avery R, Badshah C, Boeckh M, Fournier M, Hodowanec A, Komatsu T, Limaye AP, Manuel O, Natori Y, Navarro D, Pikis A, Razonable RR, Westman G, Miller V, Griffiths PD, Kotton CN; CMV Definitions Working Group of the Transplant Associated Virus Infections Forum. Consensus Definitions of Cytomegalovirus (CMV) Infection and Disease in Transplant Patients Including Resistant and Refractory CMV for Use in Clinical Trials: 2024 Update From the Transplant Associated Virus Infections Forum. Clin Infect Dis. 2024 Sep 26;79(3):787-794. doi: 10.1093/cid/ciae321. PMID 39041385